CLINICAL TRIAL: NCT05426252
Title: Thal-FabS: Novel Transplant Strategy for High-risk Thalassemia Patients - a Phase I/II Trial of Early Fludarabine Followed by Abatacept and Sirolimus Immunosuppression
Brief Title: Thal-Fabs: Reduced Toxicity Conditioning for High Risk Thalassemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Thalassemia Foundation of Canada (Unknown)
Responsible Party: Principal Investigator, Yogi Chopra, Staff Physician, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000075672
Record Dates: First submitted 2022-06-11; First posted 2022-06-21 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Thalassemia in Children
Keywords: thalassemia; reduced toxicity; abatacept; sirolimus; pre transplant immunosuppression
MeSH Terms: conditions — Thalassemia | interventions — Abatacept; Sirolimus

STUDY DESIGN:
Intervention Model Description: Single arm, non-randomized phase I/II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PTIS followed by abatacept and sirolimus (Experimental): Administration of reduced-toxicity conditioning regimen combined with pre-transplant immunosuppression, followed by abatacept and sirolimus as graft-versus-host disease (GVHD) prophylaxis for allogeneic transplant with either Human Leukocyte Antigen (HLA)-matched sibling donors or haploidentical donors
  Interventions: Drug: Abatacept; Drug: Sirolimus

INTERVENTIONS:
Drug: Abatacept — Abatacept, co-stimulation blockade, to be given for GVHD prophylaxis in combination with sirolimus post allogeneic hematopoietic stem cell transplantation.
  Other Names: Orencia
Drug: Sirolimus — Sirolimus, mTOR inhibitor, to be given for GVHD prophylaxis in combination with abatacept post allogeneic hematopoietic stem cell transplantation.
  Other Names: Rapamicin

SUMMARY:
The purpose of this study is to evaluate a novel transplant strategy for the long-term benefit of patients with transfusion dependent high-risk thalassemia.

DETAILED DESCRIPTION:
Patients with high-risk thalassemia meeting the eligibility criteria for this study will be entered sequentially until completion or closure of the study.

The hypothesis is that a reduced-toxicity conditioning regimen combined with pre-transplant immunosuppression, followed by abatacept and sirolimus as graft-versus-host disease (GVHD) prophylaxis for allogeneic transplant with either Human Leukocyte Antigen (HLA)-matched sibling donors or haploidentical donors is feasible and safe and can be delivered with less toxicity, durable donor engraftment, and minimal GVHD.

ELIGIBILITY:
Inclusion Criteria: In order to be eligible to participate in this study, the recipient must meet all of the following criteria:

1. Patients with a diagnosis of transfusion dependent beta or alpha thalassemia (3 or 4 gene deletion) between the age of 1-18 years.
2. Thalassemia genotype must be confirmed by molecular genetic testing.
3. Patients with thalassemia must have at least one of the high-risk features:

   * Age >7 years
   * Hepatomegaly (2 cm below costal margin)
   * Inadequate iron chelation (liver iron content >7mg/g dry weight)
   * Severe alloimmunization
   * Unable to tolerate iron chelation

3. Patients must have had a complete evaluation of their iron status including measurement of serum ferritin, MRI of the heart and liver (within the previous 6 months prior to referral). Liver elastography (within the preceding 3 months) will be also obtained but not required.

4. Ability to take oral medication and be willing to adhere to the study regimen.

5. Patients who have a performance status of at least 70% Karnofsky or Lansky status prior to transplantation.

6. Patients who are acceptable candidates for marrow transplantation based on their pre-BMT evaluation.

7. Patients who have histocompatibility sibling or HLA haplo identical family member and have been medically approved as hematopoietic progenitor cell donors.

8. Patients who are not candidates for gene therapy.

9. Patients/legal guardians who sign informed consent for the protocol approved by the Research Ethical Board of the Hospital for Sick Children/University of Toronto.

Exclusion Criteria: The recipient who meets any of the following criteria will be excluded from participation in this study:

1. Patients will not be excluded based on sex, race, or ethnic background.
2. Patients will be excluded if they demonstrate significant functional deficits in major organs, which could interfere with the outcome following bone marrow transplant, including:

   * Cardiac: Evidence of significant cardiac dysfunction (resting left ventricular ejection fraction of < 50% with absence of improvement with exercise), marked cardiomegaly or uncontrollable hypertension.
   * Renal: Evidence of > 50% reduction in expected creatinine clearance or GFR < 60mL/min/1.73m2
   * Hepatic: Evidence of hepatic dysfunction evidenced by a serum direct (conjugate) bilirubin of > 2.5 mg/dl, or ALT > 5 times the upper limit of normal for age.
   * Pulmonary: Evidence of focal or diffuse active infection or pneumonitis and the patient demonstrates a FEV1 < 50% or carbon monoxide diffusing capacity (DLCO) of < 50% predicted value (adjusted for hemoglobin). The patient should not require ventilation support.
3. Presence of donor specific antibody (DSA) with mean fluorescence intensity (MFI) greater than 3,000.
4. Previous stem cell transplant or gene therapy.
5. Presence of cardiomyopathy with a T2* < 10ms per Cardiac MRI.
6. Presence of significant liver iron deposition defined as liver iron content >15mg/g liver dry weight. If iron chelation were optimized and reassessment within 6 months shows a decrease of LIC to <15 with no evidence of cardiomyopathy, patient may still be considered for enrollment.
7. Active HIV, hepatitis B or hepatitis C disease.
8. Severe liver cirrhosis or bridging fibrosis on liver biopsy if previously done.
9. Prior or current malignancy or myeloproliferative or immunodeficiency disorder.
10. Evidence of active, deep seated, life-threatening infections despite therapy (e.g., certain fungal species, HIV, etc.).
11. Patients will be excluded if they are women of childbearing potential who are currently pregnant (b-HCG+) or who are not practicing adequate contraception.
12. Any condition that would preclude serial follow up.
13. Patients with a known life-threatening allergy to components of the pre transplant immunosuppression (fludarabine), conditioning (treosulfan, cyclophosphamide or anti-thymocyte globulin) or graft versus host prophylactic regimen (abatacept, sirolimus).
14. Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk

Donor Eligibility:

Donors will not be considered research subjects as the stem cell collection procedure is standard of care and will not be considered part of the research.

In order to be eligible to participate in this study, the donor must meet all of the following criteria:

1. May have thalassemia or sickle trait.
2. Will also consider ABO match and lack of donor specific anti-HLA antibodies.
3. Donors must be minimal of 15 kg weight and have completed routine donor evaluations as per our standard of care.
4. Donors must have signed (by patient or legal guardian) informed consent for the protocol approved by the Research Ethical Board of the Hospital for Sick Children/University of Toronto.
5. No evidence of transmissible diseases in compliance with the Health Canada CTO regulations
6. Not pregnant or lactating
7. Must not be allergic to granulocyte colony stimulating factor (G-CSF)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have WBC engraftment by day +100 | Until Day +100
  Rate of neutrophil engraftment defined by the first day of 3 consecutive days of absolute neutrophil counts above 500/uL after bone marrow transplant.
Number of patients who develop Grade II to IV acute GVHD at Day +100 | Until Day +100
  Incidence of Grade II or greater acute graft-versus-host disease (GvHD) post-transplant using criteria by Przepiorka et al, 1994
Immune reconstitution | Until Day +365
  Rate of immune reconstitution defined by recovery of CD4 cells post bone marrow transplantation

SECONDARY OUTCOMES:
Number of patients who develop Chronic GVHD | Day +100 until Day +365
  Incidence of chronic GVHD using NIH consensus staging system at 6 months and 1 year

OTHER OUTCOMES:
Number of patients who will wean Sirolimus at 1 year post transplant | Until Day +365
  Numbers of patients eligible to wean sirolimus at 1 year.
Length of stay | Until Day +365
  Numbers of length of hospital stay after bone marrow transplant
Cost effectiveness | Until Day +365
  Amount of cost including utilization of healthcare throughout transplant

CONTACTS AND LOCATIONS:
Overall Officials: Yogi Chopra, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Yogi Chopra, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raffa EH, Harris TM, Choed-Amphai C, Kirby-Allen M, Odame I, Ali M, Krueger J, Hermans KG, Tole S, Seelisch J, Klaassen RJ, Abbott L, Chopra YR, Wall DA, Chiang KY. Early Engraftment and Immune Kinetics Following Allogeneic Transplant Using a Novel Reduced-Toxicity Transplant Strategy in Children/Adolescents with High-Risk Transfusion-Dependent Thalassemia: Early Results of the ThalFAbS Trial. Transplant Cell Ther. 2025 Mar;31(3):180.e1-180.e12. doi: 10.1016/j.jtct.2024.12.016. Epub 2024 Dec 24. PMID 39722321